CLINICAL TRIAL: NCT02360098
Title: Determinants of the Pattern of Emergence From Anesthesia in Patients Undergoing Anterior Temporal Lobectomy and Amygdalohippocampectomy
Brief Title: Emergence From Anesthesia in Anterior Temporal Lobectomy and Amygdalohippocampectomy Patients
Status: Completed | Type: Observational
Sponsor: Lashmi Venkatraghavan (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Sponsor-Investigator, Lashmi Venkatraghavan, Assistant Professor, Department of Anesthesia, Toronto Western Hospital, Toronto, Canada, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Other Study IDs: UHN REB 14-8212 BE
Record Dates: First submitted 2015-02-02; First posted 2015-02-10 (Estimated); Results first posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Emergence From Anesthesia
Keywords: Emergence from Anesthesia; Anterior temporal lobectomy; Amygdalohippocampectomy; Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Emergence from Anesthesia — There are no study related interventions in this study and perioperative care of these patients will be as per our standard practice The only study related protocol would be collecting the data on the emergence from anesthesia. The data will be collected from the time of turning off the anesthetic agents till the discharge from recovery room. Data collected include, vital signs, Glasgow coma scale( GCS), and Riker agitation- sedation score.. The patients will be assessed every 5 minutes for the first 30 minutes and every 10 minutes for the next 60 minutes.

SUMMARY:
Smooth emergence (wake up) from anesthesia is an important consideration in patients undergoing neurosurgical procedures as blood pressure changes associated with violent emergence can cause intracranial hemorrhage and brain swelling. At the same time, emergence should also be quick so that patients' neurological function can be assessed at a timely manner. Pattern of emergence from anesthesia is poorly investigated and understood.

DETAILED DESCRIPTION:
Epilepsy surgery involves resecting epileptogenic tissues including limbic structures which may be functionally normal. Hence the emergence process can be complicated in patients having diseased limbic structures or those having therapeutic removal of limbic structures as in epilepsy surgery. Limbic structures are responsible for memory, language and executive function and hence loss of some of these higher functions is to be expected in the postoperative period. Preoperative neuropsychological assessments are often used to predict their risk for postoperative loss of higher functions and behavior changes. In our experience the investigators have seen that there is a spectrum of emergence characteristics in patients undergoing temporal lobectomy that can vary from dangerously agitated patient to much sedated, unarousable patient. Delirium and agitation can be dangerous and have serious consequences for the patient such as injury, increased pain, hemorrhage, self-extubation and removal of catheters requiring physical or chemical restraint. On the other hand the unarousable patient may pose dangerous airway complications and limit neurological assessment in the immediate postoperative period. Hence it is essential to have a clue about post anesthesia emergence behavior in patients having epilepsy surgeries. The aim of this study is to look at the pattern of emergence from anesthesia after epilepsy surgery and to determine if preoperative neuropsychological assessment help predict the pattern of emergence in patients undergoing anterior temporal lobectomy and amygdalohippocampectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients above the age of 18 who are scheduled for elective anterior temporal lobectomy and amygdalohippocampectomy under General Anesthesia

Exclusion Criteria:

* Lack of informed consent Patients needing intensive care unit postoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergence from anesthesia in anterior temporal lobectomy and amygdalohippocampectomy PATIENTS
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2014-12; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lashmi Venkatraghavan, MD, Principal Investigator — Toronto Western Hospital/UHN
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: all patients will be seen by the anesthesiologists in the pre-anesthesia consult clinic.
Pre-assignment Details: Intraoperatively, all patients will have standard monitoring consisting of electrocardiography (ECG), pulse oximetry, end-tidal carbon dioxide (ETCO2), invasive and non-invasive blood pressure, temperature, urine output, depth of anesthesia (Entropy) and end tidal anesthetic agent concentration.
Groups:
- Agitated Emergence and Smooth Emergence: Number of consented patients to participate in the study
Period: Overall Study
Arm/Group | Agitated Emergence and Smooth Emergence
Started | 36
Completed | 29
Not Completed | 7
Not completed — Physician Decision | 7

BASELINE CHARACTERISTICS:
Population: Comparison between agitated emergence and smooth emergence groups Sex/Gender data were not collected.
Groups:
- Agitated Emergence: Demographic variables of patients woke up agitated from anesthesia
- Smooth Emergence: Demographic variables of patients with smooth wake up from anesthesia
- Total: Total of all reporting groups
Arm/Group | Agitated Emergence | Smooth Emergence | Total
Number analyzed (Participants) | 9 | 20 | 29
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 33 (11) | 36 (13) | 34.5 (12)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Sex/Gender data were not collected.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Mean (Standard Deviation); unit: Kg] | 76 (15) | 75 (19) | 75.5 (17)
Height [Mean (Standard Deviation); unit: cm] | 174 (10) | 170 (9) | 172 (8)

OUTCOME MEASURES:

1. Primary Outcome: Volumes of the Hippocampus, Thalamus and Amygdala
Description: Comparison of volumes of the hippocampus, thalamus and amygdala between Agitated and Smooth emergence groups
Time Frame: 1 day
Population: Comparison of volumes of the hippocampus, thalamus and amygdala in both groups
Measure: Mean (Standard Deviation); unit: mm3
Groups:
- Agitated Emergence; Smooth Emergence: Comparison of volumes of the hippocampus, thalamus and amygdala
Arm/Group | Agitated Emergence | Smooth Emergence
Number analyzed (Participants) | 9 | 20
mm3
  ipsilateral hippocampus | 3578 (344) | 3903 (516)
  contralateral hippocampus | 3479 (452) | 3525 (569)
  ipsilateral thalamus | 7311 (663) | 7479 (856)
  contralatera thalamus l | 7608 (908) | 7631 (799)
  ipsilateral amygdala | 1331 (272) | 1295 (285)
  contralateral amygdala | 1321 (223) | 1260 (230)

ADVERSE EVENTS:
Time Frame: 1 day
Description: Any adverse events detected.
Groups:
- Agitated Emergence and Smooth Emergence: Demographic variables and anesthetic agent use
Arm/Group | Agitated Emergence and Smooth Emergence
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT02360098/Prot_SAP_000.pdf